CLINICAL TRIAL: NCT00352092
Title: A Pilot Study of Corticosteroid-Free, Calcineurin-Sparing Immunosuppression Protocol for HLA-Identical Living Donor Renal Transplant Recipient
Brief Title: Pilot Study for HLA Identical Living Donor Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Rita Alloway, Research Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEL313
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Renal Transplant
Keywords: Kidney disease; Renal transplant; HLA Identical; Living Donor; Corticosteroid free; Calcineurin sparing; Adults
MeSH Terms: conditions — Kidney Diseases | interventions — Calcineurin Inhibitors; Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: calcineurin inhibitor
Drug: sirolimus
Drug: mycophenolate mofetil

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of a steroid-free and calcineurin-inhibitor free treatment regimen for patients who are receiving a kidney transplant from a living donor that is HLA-identical (has a similar immune system).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and effectiveness of a steroid-free and calcineurin-inhibitor free treatment regimen for patients who are receiving a kidney transplant from a living donor that is HLA - identical, or in other words, has a similar immune system. The immune system is a defense system that the body uses to fight foreign substances that enter the body, such as a transplanted kidney. Two people with similar immune systems are less likely to fight off or reject an organ donated from one to the other. HLA-identical kidney transplant recipients are less likely to need large amounts of immunosuppression because they are immunologically similar. In this study, you will be treated with the immunosuppressive medications, Cellcept, Rapamune, and Prograf and after a rejection free period will remain on Cellcept alone. This treatment regimen is currently being used at The University of Cincinnati for all HLA-identical living donor kidney transplant recipients. This study is being conducted to determine if the protocol currently being used results in beneficial outcomes for HLA-identical kidney transplant recipients.

Only recently have transplant centers considered avoiding steroid therapy (prednisone) in any transplant patient because steroids have been used successfully for so long, but with many side effects. The ability to stop steroids has occurred due to the availability of newer more effective immunosuppressive medications. Stopping steroids has been tried in patients who are considered to be at both low and higher risk of kidney rejection. Patients considered at risk for rejection may typically be left on steroids forever or no attempts to stop the steroids would be made until the patient is one year after transplant and has already received a lot of steroid therapy resulting in side effects. This study will be conducted in patients that are low risk for rejection and can potentially benefit from steroid avoidance.

Overall, the concept of steroid avoidance in patients that are at low risk for rejection is now much more acceptable because newer, more potent medications have recently become available to prevent acute rejection. These newer medications include Prograf (tacrolimus), Cellcept (mycophenolate mofetil), and Rapamune (sirolimus). Currently, most kidney transplant recipients receive medications consisting of tacrolimus or cyclosporine, mycophenolate mofetil or azathioprine, and steroids. However, recently, the combination of Prograf (tacrolimus) and Rapamune (sirolimus) with steroid withdrawal 3 months after transplantation was studied in patients receiving liver, liver/kidney, and kidney/pancreas transplants. This study showed a low rate of acute rejection with excellent patient and kidney survival.

The addition of Cellcept to Prograf and Rapamune is thought to be a safe and effective alternative to the use of steroids in transplant patients. Due to the low risk of rejection for HLA-identical kidney transplant recipients, patients in this study will be slowly withdrawn from both Rapamune and Prograf over a rejection free period of time. Withdrawal of these medications and avoidance of steroids could decrease the development of high blood pressure, high cholesterol, diabetes, tremors, and infection after transplant. This study will determine if this medication regimen is safe, effective, and able to produce beneficial post transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Male/female recipients
* All ethnic groups
* Negative pregnancy test
* Practicing an acceptable form of birth control
* Signing informed consent

Exclusion Criteria:

* Known sensitivity or contraindication to mycophenolate mofetil, tacrolimus, or sirolimus
* Re-transplants who lost primary transplant from immunologic causes (patients with graft loss secondary to technical or calcineurin-inhibitor toxicity will be included)
* Liver, heart, pancreas or small bowel transplant recipient
* Fasting total cholesterol >300 mg/dL and fasting triglycerides >400 mg/dL
* Baseline WBC count <3000/cu.mm
* Baseline platelet count <100,000/cu.mm
* Known or suspected malignancy within previous 3 years, (Patients with squamous cell and basal skin cancer are not excluded)
* Active systemic infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy confirmed acute rejection at 12 and 24 months.

SECONDARY OUTCOMES:
Patient survival
Graft survival
Early discontinuation of mycophenolate mofetil, tacrolimus, or sirolimus due to toxicity
Time to acute rejection from transplant
Severity of acute rejection measure by Banff'93 criteria, and/or requirement of antilymphocyte treatment; need for corticosteroid pulse or maintenance therapy for rejection or recurrent disease
Evaluation of 24-hour proteinuria at 24 months post-transplant
Evaluation of graft function by calculated CrCl (Cockroft-Gault) at 1, 3, 6, 12, and 24 months post-transplant
Patient weight
Quantitative bone loss
Cholesterol and triglyceride levels at 12 and 24 months
Cardiovascular risk assessment by Framingham criteria at 0, 1, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rita Alloway, Pharm.D., Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States